CLINICAL TRIAL: NCT01088581
Title: Adjuvant Hepatic Arterial Infusional Chemotherapy With 5-fluorouracil and Cisplatin After Curative Resection of Hepatocellular Carcinoma: A Prospective Randomized Study
Brief Title: Adjuvant Hepatic Arterial Infusional Chemotherapy After Curative Resection of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2005-0203
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatic arterial infusion chemotherapy; 5-fluorouracil; cisplatin; adjuvant chemotherapy; hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation group (No Intervention): No adjuvant chemotherapy after resection
- Adjuvant group (Active Comparator): Adjuvant chemotherapy after resection
  Interventions: Drug: Adjuvant group

INTERVENTIONS:
Drug: Adjuvant group — Adjuvant chemotherapy (5FU and cisplatin) after resection
  Other Names: Adjuvant chemotherapy after resection
  Arms: Adjuvant group

SUMMARY:
Several adjuvant therapies have been attempted to reduce uni-centric, and intra- or extrahepatic recurrence after curative surgical resection for hepatocellular carcinoma (HCC). However, because the efficacy of such adjuvant therapy remains unclear, there is no standard postoperative therapy.

The investigators investigated whether adjuvant hepatic arterial infusional chemotherapy with 5-fluorouracil (5-FU) and cisplatin reduces the recurrence of HCC after curative resection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignancies in the world. In particular, the global occurrence rate of HCC ranks first in males and fourth in females. Despite advances in diagnosis and medical, and surgical management, HCC is still considered a difficult disease to cure because of the high recurrence rate, even after surgical resection. The cumulative 3-year recurrence rate after resection with a curative aim is approximately 80%.1 Portal vein invasion and satellite nodules are important factors that predispose a patient to recurrence after resection.2 More importantly, recurrence after resection usually results in a high rate of mortality.3 Uni-centric or intrahepatic metastatic recurrence usually indicates metastatic spread from the primary tumor and is generally distinguished from multi-centric recurrence by a short interval between resection and recurrence (12 months for primary tumor spreading vs. 3 years for multi-centric recurrence).4,5 In this regard, several adjuvant therapies have been used to attempt to primarily reduce uni-centric, and intra- or extrahepatic recurrence after curative surgical resection for HCC. However, because the efficacy of adjuvant therapy after curative resection is still not clear, no recommendation for postoperative therapy exists.

Several chemotherapeutic agents, including doxorubicin, epirubicin, mitomycin C, 5-fluorouracil (5-FU), and cisplatin have been delivered into the hepatic artery via an implanted port system as the first-line regimen or adjuvant therapy after curative resection in HCC.6-8 A recent study reported that repetitive short-course hepatic arterial infusion of 5-FU and cisplatin showed significant anti-tumor effects in advanced HCC.9 With the hypothesis that post-operative chemotherapeutic agents delivered via the hepatic artery may eliminate residual cancer cells in the liver, we designed a prospective study to determine whether adjuvant hepatic arterial infusional chemotherapy (HAIC) with 5-FU and cisplatin reduced the incidence of recurrence of HCC and improved overall patient survival after curative resection.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 to 70 years old
* appropriate blood test results (white blood cells (WBCs) ≥3,000/mm3, platelet count ≥50,000/mm3, total bilirubin <3mg/dl)
* a patient could enter this study if one of the following was fulfilled

  1. maximum diameter of HCC ≥5 cm,
  2. microvascular or bile duct invasion upon pathological examination,
  3. capsular invasion of HCC upon pathological examination, 4) Edmonson-Steiner grade III or IV.

Exclusion Criteria:

* patients with intra- or extrahepatic metastases at 4 weeks after resection
* Child-Pugh class B or C (n = 4)
* ECOG performance scale ≥2
* prior systemic chemotherapy, radiation, or locoregional therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
2-year recurrence rate and adverse events | 2-year

SECONDARY OUTCOMES:
overall survival | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Seung Up Kim, MD, Study Director — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea